CLINICAL TRIAL: NCT07263971
Title: Birth Experiences of Women Giving Birth in French-speaking Belgium and Pathways to Choosing a Place of Birth
Brief Title: Birth Experience of Women Giving Birth in Belgium
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: NAISSANCE
Record Dates: First submitted 2025-09-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related
Keywords: Birthplace Choice; Birth Experience

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women who have given birth: Qualitative interviews with women who have given birth
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Other: Qualitative Interview — Qualitative interview with volunteering women having given birth.

SUMMARY:
The aim of this research is to understand what motivates women giving birth in Belgium to choose a particular place of birth and their experiences of childbirth. This understanding is made possible by collecting qualitative data from women who have given birth (from the first month after giving birth up to one year postpartum). The objective here is to understand what motivates the choice of place of birth (with a focus on the notion of 'non-choice') and to gain insight into the childbirth experiences of women giving birth in Belgium. The researcher also meets with birth companions (perinatal health professionals and birth companions such as doulas, for example) to understand their professional practice and their choice of workplace (home, birth centre or cottage, traditional hospital ward, university hospital ward, etc.).

ELIGIBILITY:
Inclusion Criteria:

* have given birth in Belgium
* have given birth less than a year ago
* be of legal age
* volunteer

Exclusion Criteria:

* not having given birth once in Belgium
* being a minor

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women having given birth within a year
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Birth experience | Throughout the entire study, approximately during 40 months
  The outcome is how women have experience their delivery. As it is through qualitative interviews, we can not yet specify the results.
Birthplace Choice | Throughout the entire study, approximately during 40 months
  Which birthplace women have choosen, do they have the feeling they had a choice. If yes : how women choose the birth place, when and what influenced them in their decision. If not : who took the decision and why.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain, Brussels, Woluwe-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: No